CLINICAL TRIAL: NCT05213377
Title: Effect of Preoperative Warming on Intraoperative Hypothermia and Postoperative Functional Recovery Outcomes in Direct Anterior-approached Total Hip Arthroplasty: a Randomized Clinical Trial
Brief Title: Preoperative Warming, Hypothermia and Functional Recovery in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Michele Carella, Head of Clinic, Anesthesiology and Intensive Care Department, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Thermo-ATHA22
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Hypothermia Following Anesthesia; Hypothermia; Anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (No Intervention): Patients undergoing total hip replacement surgery by anterior approach, with general anesthesia and continuous core body temperature measurement via nasopharyngeal thermic probe.
  Patients recruited for surgery who will not receive the 30 minutes of preoperative warming through pulsed air thermal coverage.
- Group W (Experimental): Patients undergoing total hip replacement surgery by anterior approach, with general anesthesia and continuous core body temperature measurement via nasopharyngeal thermic probe.
  Patients recruited for surgery who will receive the 30 minutes of preoperative warming through pulsed air thermal coverage.
  Interventions: Procedure: Preoperative warming

INTERVENTIONS:
Procedure: Preoperative warming — Patients enrolled in surgery who will not receive 30 minutes of pulsed air thermal blanket warming prior to induction of anesthesia (3M™ Bair Hugger™ Adult Integral Blanket, Model 300 Dimensions: 213 cm x 91 cm)
  Arms: Group W

SUMMARY:
This prospective, randomized, single-center study compares intraoperative heat loss at the core temperature level in patients scheduled for direct anterior total hip arthroplasty under general anesthesia and who will or will not, according to randomization, receive one hour of pre-warming with a pulsed air thermal blanket prior to anesthesia induction.

DETAILED DESCRIPTION:
In patients undergoing surgery, intraoperative hypothermia can occur because of anesthesia-induced inhibition of thermoregulation and heat loss associated with the patient's exposure to an environment maintained at a temperature below normal skin temperature.

Randomized trials show that even mild hypothermia results in serious complications, including surgical wound infection, coagulopathy and increased blood transfusions, and delayed postoperative recovery.

All products used during general anesthesia profoundly alter thermoregulatory control, reducing the activation thresholds of the main defenses against cold, which are the closure of the arteriovenous shunt and the generation of shivering. Impaired thermoregulation, combined with a cold operating room environment and direct-anterior hip surgical approach and exposure, causes hypothermia in almost all unheated patients.

The body core temperature is finely tuned to maintain an average of 37°C by balancing heat gain and loss. The nasopharynx is an excellent alternative to patient core temperature monitoring when esophageal monitoring is excluded for surgical reasons or blocked by an airway protected by an airway device.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3
* Scheduled for direct anterior-approached total hip replacement surgery under general anesthesia

Exclusion Criteria:

* pregnant women
* patients with:

  1. peripheral neuropathy or other severe neurological pathology
  2. immunosuppression
  3. chronic renal insufficiency or severe hepatic insufficiency
  4. major congenital or acquired hemostasis disorders
  5. craniofacial dysmorphism or anatomical alterations of the upper airways
  6. known thermoregulatory disorders
* patients with a preoperative body temperature > 37.5°C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Core body temperature | Intraoperative
  Variation of core body temperature during surgery, i.e. the difference between the temperature at the time of induction of general anaesthesia and the minimum temperature recorded during the procedure, as well as its evolution over time.

SECONDARY OUTCOMES:
Intraoperative blood loss | Intraoperative
  Total intraoperative blood loss
Shivering | First 6 hours after surgery
  The incidence of shivering in the first 6 hours post-surgery
Patient comfort | First 6 hours after surgery
  Comfort in the recovery room by visual analogical scale (VAS 0-100)
Patient comfort | First 6 hours after surgery
  Length of stay in the recovery room
Surgical site infection | 30 days after surgery
  Incidence of surgical site infection at 30 days postoperative
Postoperative complications | 3 days after surgery
  The occurrence of side effects related to hypothermia (cardiovascular, infectious and hemorrhagic complications)
QoR-15 | Day-1 and Day-3 after surgery
  Postoperative patient satisfaction and functional outcome (QoR-15 at D1 and D3)
LoS | 30 days after surgery
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Simpson JB, Thomas VS, Ismaily SK, Muradov PI, Noble PC, Incavo SJ. Hypothermia in Total Joint Arthroplasty: A Wake-Up Call. J Arthroplasty. 2018 Apr;33(4):1012-1018. doi: 10.1016/j.arth.2017.10.057. Epub 2017 Nov 8. PMID 29195854
- [Background] Akca O, Sessler DI. Thermal management and blood loss during hip arthroplasty. Minerva Anestesiol. 2002 Apr;68(4):182-5. PMID 12024079
- [Background] McClain R, Bojaxhi E, Ford S, Hex K, Whalen J, Robards C. Forced-Air Convection Versus Underbody Conduction Warming Strategies to Maintain Perioperative Normothermia in Patients Undergoing Total Joint Arthroplasty. Cureus. 2020 Nov 13;12(11):e11474. doi: 10.7759/cureus.11474. PMID 33329970